CLINICAL TRIAL: NCT03816514
Title: Use of Noninvasive Hemoglobin Monitoring for Maintaining Hemoglobin Concentration Within the Target Range During Major Surgery: A Randomized Controlled Trial
Brief Title: Noninvasive Hemoglobin Monitoring for Maintaining Hemoglobin Concentration Within the Target Range
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-1811-039-986
Record Dates: First submitted 2018-12-17; First posted 2019-01-25 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Hemoglobins; Blood Transfusion; Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpHb monitoring group (Experimental): In SpHb monitoring group, noninvasive, continuous SpHb monitoring will be done using Radical-7 pulse CO-Oximeter. The patients will be managed according to the prespecified protocol based on the SpHb values.
  Interventions: Procedure: SpHb monitoring
- Control group (Active Comparator): In control group, patients will receive conventional management without the SpHb monitoring. In these patients, the information about hemoglobin concentration of the patients will be obtained from hemoglobin measurement analyzed by point-of-care (POC) equipment, as usual standard care.
  Interventions: Procedure: Conventional management

INTERVENTIONS:
Procedure: SpHb monitoring — Noninvasive, continuous pulse oximetry-based hemoglobin (SpHb) monitoring
  Arms: SpHb monitoring group
Procedure: Conventional management — Conventional management without SpHb monitoring
  Arms: Control group

SUMMARY:
The primary aim of this study is to evaluate whether pulse oximetry based noninvasive hemoglobin (SpHb) monitoring can reduce the incidence of hemoglobin (Hb) level out of the target range in adult patients undergoing major surgery with the potential risk of bleeding.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ASA physical status class I, II, III, who scheduled to undergo elective non-cardiac major surgery with more than moderate risk of bleeding under general anesthesia or spinal anesthesia.
* Eligible Surgery include: Spine surgery, bone tumor surgery, Total Hip Replacement, ovarian cancer surgery, cervical cancer surgery, radical cystectomy, open retroperitoneal mass excision, Radical Retropubic Prostatectomy, explorative laparotomy for abdominal mass excision, abdominal aortic aneurysm repair
* Patients who are requiring an arterial catheter as a part of their standard care.

Exclusion Criteria:

* Patients with preexisting deformity or skin condition that would impede sensor placement
* Patients with allergies to the adhesive sensor material
* Patients with uncorrected preoperative anemia (preoperative hemoglobin < 7 g/dL)
* Patients who were not suitable for participation in the opinion of the study investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-11-02 (Actual); Study Completion 2020-11-06 (Actual)

PRIMARY OUTCOMES:
The incidence of deviation from the target hemoglobin range | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  (The number of laboratory samples with the result hemoglobin concentrations were out of the target range)/(Total number of laboratory samples that performed during intra-operative periods)

SECONDARY OUTCOMES:
The percentage extent of deviation from the target hemoglobin range | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  The percentage extent of deviation of laboratory hemoglobin out of the prespecified target range
Number of Point-of-care (POC) sampling during surgery | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Number of Point-of-care (POC) sampling for measurement of hemoglobin concentration. In SpHb group, POC sampling will be done according to SpHb level. In control group, POC sampling will be done at discretion of anesthesiologist.
Accuracy of the SpHb value | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Standard Laboratory hemoglobin measurement will be used as reference. Laboratory measurements will be done every 30 minute during surgery
Number of patients who receive intra-operative transfusion | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Number of patients who were transfused with pRBCs intraoperatively
Total volume of intravenous fluids given | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Total volume of intravenous fluids given intra-operatively
Total volume of pRBCs transfused | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Total volume of pRBCs transfused intra-operatively
Time for transfusion delay | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  Time from the determination of transfusion to actual transfusion, in minutes
Incidence of intraoperative hypotension | Until transfer to PACU (Post-Anesthesia Care Unit), from the beginning of the induction of anesthesia
  hypotension is defined as SBP < 80% of baseline SBP
laboratory total hemoglobin value, at postoperative day 1 | at postoperative day 1
  total hemoglobin value measured by standard laboratory method

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul national university hospital, Seoul, South Korea

REFERENCES:
- [Background] Berkow L, Rotolo S, Mirski E. Continuous noninvasive hemoglobin monitoring during complex spine surgery. Anesth Analg. 2011 Dec;113(6):1396-402. doi: 10.1213/ANE.0b013e318230b425. Epub 2011 Sep 29. PMID 21965372
- [Background] Causey MW, Miller S, Foster A, Beekley A, Zenger D, Martin M. Validation of noninvasive hemoglobin measurements using the Masimo Radical-7 SpHb Station. Am J Surg. 2011 May;201(5):592-8. doi: 10.1016/j.amjsurg.2011.01.020. PMID 21545905
- [Background] Galvagno SM Jr, Hu P, Yang S, Gao C, Hanna D, Shackelford S, Mackenzie C. Accuracy of continuous noninvasive hemoglobin monitoring for the prediction of blood transfusions in trauma patients. J Clin Monit Comput. 2015 Dec;29(6):815-21. doi: 10.1007/s10877-015-9671-1. Epub 2015 Mar 10. PMID 25753142
- [Derived] Park SK, Hur C, Kim YW, Yoo S, Lim YJ, Kim JT. Noninvasive hemoglobin monitoring for maintaining hemoglobin concentration within the target range during major noncardiac surgery: A randomized controlled trial. J Clin Anesth. 2024 May;93:111326. doi: 10.1016/j.jclinane.2023.111326. Epub 2023 Nov 20. PMID 37988814